CLINICAL TRIAL: NCT06686524
Title: Clinical Study of CD19 Targeted Universal Chimeric Antigen Receptor T Lymphocytes (UCAR-T) for the Treatment of Refractory Juvenile Dermatomyositis (RJDM)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC081
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Dermatomyositis, Juvenile; Dermatomyositis
Keywords: Dermatomyositis; CD19; UCAR-T; Universal CAR-T
MeSH Terms: conditions — Dermatomyositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anti-CD19 UCAR-T cells (Experimental)
  Interventions: Drug: Anti-CD19 UCAR-T cells

INTERVENTIONS:
Drug: Anti-CD19 UCAR-T cells — A single infusion of CD19 UCAR-T cells will be administered intravenously after lymphodepletion chemotherapy.

SUMMARY:
This study is an open-label, single-arm, dose-escalation trial primarily designed to evaluate the safety and efficacy of a universal CAR-T cell therapy targeting CD19 in the treatment of patients with RJDM. Additionally, the study aims to characterize its pharmacokinetic and pharmacodynamic properties, explore its role in immune system reconstitution, and assess long-term survival benefits.

DETAILED DESCRIPTION:
This study adopts the "3+3" design, with a total of three dosage groups (1 × 107/kg, 3 × 107/kg, 6 × 107/kg). The study will start from the low dose group. Only when the present dose group has completed enrollment and no DLT has been observed, the study could escalate to the next dose group based on the evaluation of efficacy and cell kinetic data. If no DLT is observed even in the highest dose group, the escalation will be terminated.Each dose group is expected to enroll 3 to 6 patients, with a total of 9 to 18 patients anticipated in the trial.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥ 5 years old;
* (2) Diagnosis of juvenile dermatomyositis (JDM) according to Bohan and Peter criteria;
* (3) Meeting the classification criteria for RJDM, and meeting condition ① and any one of ② to ⑤ conditions:

  * Intolerance or inadequate response to glucocorticoids (prednisone 1-2mg/kg/d or equivalent dose of other hormones) and at least two immunosuppressants, with hormone therapy lasting for at least 6 months;

    * Rapid progression of the disease and/or involvement of organs such as lungs, heart, and gastrointestinal tract;

      * Calcification of subcutaneous or muscular and articular tissues;

        * Repeated skin rashes or ulcers;

          * Repeated or persistent muscle weakness (muscle magnetic resonance imaging indicating widespread, diffuse edema or a Children's Myositis Assessment Scale (CMAS) score < 48, and at least two abnormal results among the following five core measurement indicators: Physician's Global Assessment (PhGA) ≥ 2cm, Patient's Global Assessment (PtGA) ≥ 2cm, Disease Activity Score (DAS) ≥ 2 points, Child Health Assessment Questionnaire (C-HAQ) total score ≥ 0.25 points, and muscle enzyme level > 1.5 times the upper limit of normal (ULN));
* (4)Patients with immune-mediated necrotizing myopathy who are positive for SRP or HMGCR antibodies meet the criteria for RJDM and can be directly included;
* (5) Basic normal function of important organs:

  * Cardiac function: Left ventricular ejection fraction (LVEF) ≥55%, with no significant abnormalities observed in the electrocardiogram;

    * Renal function: eGFR ≥ 30mL/min/1.73m2;

      * Liver function: AST and ALT ≤3.0 ULN, total bilirubin ≤2.0×ULN (excluding those caused by primary diseases);

        * Pulmonary function: SpO2 ≥92%;
* (6) Female subjects of childbearing age have a negative result in the urine pregnancy test and agree to take effective contraceptive measures during the trial until one year after infusion;
* (7) The patient or their guardian agrees to participate in this clinical trial and signs an informed consent form, indicating their understanding of the purpose and procedures of the clinical trial and their willingness to participate in the study.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from this trial:

* (1) Previously received CAR-T cell therapy (except for those whose safety risks have been judged as eliminated by the investigator);
* (2) Accompanied by primary immunodeficiency disease or severe secondary immunodeficiency disease that has not been corrected;
* (3) Accompanied by severe, active, or uncontrolled infectious diseases, including but not limited to active tuberculosis, latent tuberculous infection, active viral hepatitis, etc.;
* (4) Known to have active malignant diseases or confirmed malignancies before screening (including hematological malignancies and solid tumors, except for resected and cured cutaneous basal cell carcinoma);
* (5) Suffering from congenital heart disease or having a history of acute myocardial infarction within 6 months, or severe arrhythmia (including multifocal frequent ventricular supraventricular tachycardia, ventricular tachycardia, etc.); or complicated with moderate to large pericardial effusion, severe myocarditis, etc.; or unstable vital signs requiring vasopressors to maintain blood pressure;
* (6) Accompanied by other diseases that require long-term use of glucocorticoids or immunosuppressants;
* (7) Received solid organ transplantation or hematopoietic stem cell transplantation within 3 months before screening; or presence of acute graft-versus-host disease (GVHD) of grade 2 or above within 2 weeks before screening;
* (8) Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and peripheral blood hepatitis B virus (HBV) DNA titer detection is greater than the normal reference range; or positive for hepatitis C virus (HCV) antibody and peripheral blood hepatitis C virus (HCV) RNA titer detection is greater than the normal reference range; or positive for human immunodeficiency virus (HIV) antibody; or positive for syphilis test;
* (9) Received live vaccines within 4 weeks before screening;
* (10) Positive blood pregnancy test;
* (11) Participated in other clinical trials within 3 months before enrollment;
* (12) Other conditions that the investigator considers unsuitable for participation in the study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-11-11 (Estimated); Primary Completion 2026-11-10 (Estimated); Study Completion 2027-11-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 28 dyas
  The incidence of adverse events after CAR-T cell infusion was assessed by CTCAE, version 5.0.
Total improvement score (TIS) after anti-CD19 UCAR-T cells infusion. | 6 months
  The total improvement score between 0-100 also corresponds to the degree of improvement, with higher improvement scores indicating greater improvement.
Disease Activity Score (DAS) after anti-CD19 UCAR-T cells infusion. | 6 months
  Including musculoskeletal system score and skin mucosal score, with a total score of 20 points. The higher the score, the higher the disease activity
Changes of myositis specific antibody levels and serum muscle enzyme levels after anti-CD19 UCAR-T cells infusion. | 6 months
Improvement in muscle inflammation infiltration by MRI after anti-CD19 UCAR-T cells infusion. | 6 months
Childhood Myositis Assessment Scale (CMAS) score after anti-CD19 UCAR-T cells | 6 months
  The total score is 52 points, the lower the score, the weaker the muscle strength and the more severe the disease.

SECONDARY OUTCOMES:
Cmax of anti-CD19 UCAR-T cells [Cell dynamics] | 1 month
Tmax of anti-CD19 UCAR-T cells [Cell dynamics] | 1 month
AUCs of anti-CD19 UCAR-T cells [Cell dynamics] | 1 month
Changes of myth enzyme after anti-CD19 UCAR-T cells | 1 year

OTHER OUTCOMES:
Duration of disease remission (DOR) after anti-CD19 UCAR-T cells infusion [Long-term Efficacy] | 2 years
Time to B cell recovery after anti-CD19 UCAR-T cells infusion. | 1 years

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Zhejiang University School of Medicine, Hangzhou, zhejiang, Hangzhou, Zhejiang, China